CLINICAL TRIAL: NCT05299853
Title: Effects of Robot-assisted Arm Training on Respiratory Muscle Strength, Activities of Daily Living and Quality of Life in Stroke Patients: A Single-blinded Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ishtiaq Ahmed, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/34
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Rehabilitation (Experimental)
  Interventions: Other: Robot assisted arm training
- Conventional Rehabilitation (Active Comparator)
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Robot assisted arm training — Patients will receive 30 minutes of robot-assisted arm training and 30 minutes of conventional arm rehabilitation training. Patients will undergo 30 sessions of combined therapy (robotic+conventional) for a total of 6 weeks (5 sessions/week).
  Arms: Robotic Rehabilitation
Other: Conventional rehabilitation — Patients will receive 30 sessions of conventional arm training (60 minutes/day) for a total of 6 weeks (5 sessions/week).
  Arms: Conventional Rehabilitation

SUMMARY:
Stroke is the leading neurological disease in the world that causes long-term disability. The most common cause of disability after stroke is motor impairment resulting from brain damage which ultimately cause respiratory and functional limitation. Respiratory muscle weakness including the diaphragm leads to biomechanical change in respiration which can reduce vital capacity and total lung capacity of stroke patients. The weakness of diaphragm and abdominal muscle also leads to decrease in maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) in stroke patients.

Respiratory muscle training such as inspiratory or expiratory muscle training is commonly used to improve the respiratory muscle strength and function in stroke. However, it was reported that respiration is closely related to upper limb function because the muscle of upper extremities surrounds the dorsal muscle of trunk and in order to breath, the movement of trunk is necessary, which in turn is related to the movement of the upper limbs.

ELIGIBILITY:
Inclusion Criteria:

1. 18 year and above
2. Acute and sub-acute stroke patients
3. had MIP values lower than 70% of those predicted when adjusted for age and sex,
4. had no facial palsy, aphasia, or dysarthria, which would prevent respiratory muscle strength testing
5. Ischemic or Hemorrhagic stroke
6. No medical history of respiratory or lung disease

Exclusion Criteria:

1. patients with increased intracranial pressure, uncontrolled hypertension, decompensated heart failure, unstable angina, recent myocardial infarction, complicated arrhythmias, pneumothorax, bullae/blebs in the preceding 3 months
2. Any pulmonary or lungs disease
3. Any neurological conditions other than stroke
4. Using medications that could interfere with neuromuscular control or cause drowsiness.
5. Severe cognitive function (Mini-Mental Test result <24)
6. Chronic stroke
7. Recurrent stroke, brain stem stroke, and aphasia were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-06-25 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Change of baseline maximum inspiratory pressure | Baseline, Post-intervention ( 6 weeks)
  Maximum inspiratory pressure (MIP) will be measure using a hand-held mouth pressure device. Three maximal manoeuvres will perform and the highest value record. Indirect measure of respiratory (inspiratory) muscle strength, expressed in cmH20.
Change of baseline maximum expiratory pressure | Baseline, Post-intervention ( 6 weeks)
  Maximum expiratory pressure (MEP) will be measure using a hand-held mouth pressure device. Three maximal manoeuvres will perform and the highest value record. Indirect measure of respiratory (expiratory) muscle strength, expressed in cmH20.
Change from baseline ABILHAND | Baseline, Post-intervention ( 6 weeks)
  A questionnaire to assess active function of the upper limbs with 23 activities, rated as impossible, difficult or easy. The scale is scored through Rasch analysis, providing a total score ranging from -6 to +6, with higher scores indicating a lower degree of upper extremity impairment.

SECONDARY OUTCOMES:
Change from baseline Stroke Impact Scale | Baseline, Post-intervention ( 6 weeks)
  A stroke-specific health status measure featuring 16 items capturing daily activities. This scale has 8 sub-scales, evaluating: strength, hand function, mobility, activities of daily living, emotion, memory, communication and social participation. Each is rated on a 0 to 100 range (100 corresponding to least impact of stroke). An overall score is also calculated (average of sub-scales).

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırköy Dr. Sadi Konuk Eğitim ve Araştırma Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No